CLINICAL TRIAL: NCT05198713
Title: Evaluation of Hearing Aid Benefit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-487
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental (Experimental): All participants will be fit with the study hearing aid and under go the same testing conditions.
  Interventions: Device: New hearing aid

INTERVENTIONS:
Device: New hearing aid — Participants will complete testing while using a novel hearing aid which has been fit to compensate for their hearing loss.

SUMMARY:
The present study will investigate the benefit of hearing aids for speech intelligibility (in both quiet and noisy environments) compared to the unaided condition. Participants will include adults with moderate to moderately severe hearing impairment. The participants will complete laboratory-based speech intelligibility assessments with binaural hearing aids and without hearing aids.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to moderately severe sensorineural hearing loss
* Willingness to wear custom hearing instruments during the study.
* Age-normal cognition
* Ability to attend on-site study visits.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Seitz-Paquette, AuD, Principal Investigator — Sonova AG
Locations (1):
- Phonak Audiology Research Center, Aurora, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 73 [60 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Speech Intelligibility in Quiet.
Description: Speech intelligibility for monosyllabic words presented in quiet. The words are presented at a fixed level and the percentage of words correctly repeated is calculated. A higher percentage is better. This was done in both unaided and aided conditions.
Time Frame: Day 1 and Day 15
Population: It was discovered after data collection that the equipment used in this outcome measure was not functioning properly and the dB level presented was not the dB level that was indicated on the equipment. Therefore, this data was not used and no statistical analysis was done.
Measure: Mean (Full Range); unit: percentage of correct responses
Arm/Group | Experimental
Number analyzed (Participants) | 15
percentage of correct responses
  Percent correct words repeated, in a quiet condition, unaided | 92.3 [68 to 100]
  Percent correct words repeated, aided, in a quiet condition | 90.6 [64 to 100]

2. Secondary Outcome: Speech Intelligibility in Noise, Expressed as the Signal to Noise Ratio at Which Participant Can Correctly Repeat 50% of the Words
Description: Speech intelligibility on key words for sentences presented in noise. Noise is presented at a fixed level, and the words are presented at adaptive levels, below and above the noise level. A negative number is better, because it indicates the participant can correctly repeat 50% of the words when the words are below the level of noise. This was done at baseline in the unaided condition on Day 1 of the study, and in the aided condition on Day 15.
Time Frame: Day 1 and Day 15
Population: All study participants who were fit with study devices who underwent speech in noise testing in both unaided and aided conditions.
Measure: Mean (Standard Deviation); unit: dB Signal-to-Noise Ratio
Arm/Group | Experimental
Number analyzed (Participants) | 15
dB Signal-to-Noise Ratio
  dB SNR aided condition | -9.83 (1.74)
  dB SNR unaided condition | -5.87 (2.87)
Statistical Analysis 1: Comparison: Experimental; Test type: Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 15 days
Groups:
- Experimental: All participants will be fit with the study hearing aid and under go the same testing conditions. All participants underwent unaided speech in quiet and speech in noise testing on Day 1 of study. Following a 14 day field trial, all participants completed the same tests but in the aided condition. Adverse events were monitored for all participants during this two week period.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT05198713/Prot_SAP_000.pdf